CLINICAL TRIAL: NCT02594605
Title: Investigation of the Contributions of Platelet Rich Fibrin Combined With Conventional Periodontal Flap on Periodontal Healing
Brief Title: Applied The Platelet Rich Fibrin in Chronic Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Alper KIZILDAĞ, Health Sciences Institute, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 385/2012
Record Dates: First submitted 2015-10-15; First posted 2015-11-03 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet Rich Fibrin (Experimental): Platelet Rich Fibrin was applied with conventional flap surgery for treatment of periodontal bone loss in test group.
  Interventions: Device: Platelet Rich Fibrin
- Conventional Flap Surgery (Active Comparator): Platelet Rich Fibrin was not applied to control groups. Only conventional flap surgery was applied to control groups.
  Interventions: Device: Conventional Flap Surgery

INTERVENTIONS:
Device: Platelet Rich Fibrin — Platelet rich fibrin increases the growth factors. So it was applied for treatment of periodontal bone loss.
  Arms: Platelet Rich Fibrin
Device: Conventional Flap Surgery — Only Conventional Flap Surgery treatment the bone loss limitedly.
  Arms: Conventional Flap Surgery

SUMMARY:
Platelet rich fibrin is a second generation platelet concentration which contains various growth factors. The aim of this study is to evaluate the clinical and biochemical efficacy of PRF in subjects of chronic periodontitis in the operation of conventional periodontal flap.

DETAILED DESCRIPTION:
PRF was developed in 2001 by Choukroun in France, it was the second generation fibrin adhesive, and was used to accelerate the soft and hard tissue healing. Many studies have shown beneficial effects of PRF on osteoconductive filler material in sinus lift operations, treatment of periodontal sulcus defect and treatment of furcation defects. Also PRF contains many growth factors. PRF accelerates periodontal regeneration through the gradually excreted growth factors and contributes to the bone regeneration. In this study, the investigators evaluated the effect of PRF on growth factors and its contribution to periodontal regeneration in subjects with chronic periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CP who had pocket depth ≤ 5 mm and at least two area (grouped as Control and PRF) with horizontal bone loss after Phase I therapy

Exclusion Criteria:

* The subjects excluded in the study had history of systemic disease, were smokers, had allergy to any drug, had need for prophylaxis of antibiotic and had taken antibiotics at least 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Levels of IGF-1, VEGF, BMP-2, FGF-2 on Weekly | 4 weeks
  Change from baseline IGF-1, VEGF, BMP-2, FGF-2 levels of GCF at 1 month were measured by periopaper.

SECONDARY OUTCOMES:
Alteration of Clinical Attachment Level | 6 month
  Change from baseline Clinical Attachment Levels at 6 months were measured with periodontal probe.
Alteration of Periodontal Pocket Depth | 6 month
  Change from baseline Pocket Depth at 6 months were measured with periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Yasin ÇiÇEK, Study Chair — Adiyaman University
Locations (1):
- Alper KIZILDAĞ, Denizli, Denizli, Turkey (Türkiye)

REFERENCES:
- [Background] Bosshardt DD, Sculean A. Does periodontal tissue regeneration really work? Periodontol 2000. 2009;51:208-19. doi: 10.1111/j.1600-0757.2009.00317.x. No abstract available. PMID 19878476
- [Derived] Kizildag A, Cicek Y, Arabaci T, Kose O. The effect of leukocyte-platelet-rich fibrin on bone morphogenetic protein-2 and insulin-like growth factor-1 levels in patients with chronic periodontitis: a randomized split mouth clinical trail. Growth Factors. 2018 Dec;36(5-6):239-245. doi: 10.1080/08977194.2018.1551217. Epub 2019 Jan 9. PMID 30624092